CLINICAL TRIAL: NCT06338358
Title: In the Patient's Words: Understanding Patient Participation and Engagement in Plaque Psoriasis Clinical Trials
Brief Title: Understanding Participation Habits Among Plaque Psoriasis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 44519568
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Plaque Psoriasis
Keywords: Plaque Psoriasis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study intends to investigate the personal experiences of plaque psoriasis patients who take part in a separate clinical study including a specific medication intervention. The major focus will be on closely following individuals' rates of trial completion and withdrawal.

The data collected from this study will help improve future outcomes for all plaque psoriasis as well as those in under-represented demographic groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with plaque psoriasis
* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Subjects willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examination.

Exclusion Criteria:

* Refusal of consent
* Women of childbearing potential without a negative pregnancy test; or women who are lactating.
* Any serious and/or unstable pre-existing medical disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with plaque psoriasis who are actively considering enrolling in a clinical trial for said condition, but have not yet completed enrollment and randomization phases.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a plaque psoriasis clinical research. | 3 months
Number of plaque psoriasis study participants who remain in clinical study until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Armstrong AW, Gooderham M, Warren RB, Papp KA, Strober B, Thaci D, Morita A, Szepietowski JC, Imafuku S, Colston E, Throup J, Kundu S, Schoenfeld S, Linaberry M, Banerjee S, Blauvelt A. Deucravacitinib versus placebo and apremilast in moderate to severe plaque psoriasis: Efficacy and safety results from the 52-week, randomized, double-blinded, placebo-controlled phase 3 POETYK PSO-1 trial. J Am Acad Dermatol. 2023 Jan;88(1):29-39. doi: 10.1016/j.jaad.2022.07.002. Epub 2022 Jul 9. PMID 35820547
- [Background] Armstrong AW, Puig L, Joshi A, Skup M, Williams D, Li J, Betts KA, Augustin M. Comparison of Biologics and Oral Treatments for Plaque Psoriasis: A Meta-analysis. JAMA Dermatol. 2020 Mar 1;156(3):258-269. doi: 10.1001/jamadermatol.2019.4029. PMID 32022825
- [Background] Gordon KB, Langley RG, Warren RB, Okubo Y, Stein Gold L, Merola JF, Peterson L, Wixted K, Cross N, Deherder D, Thaci D. Bimekizumab Safety in Patients With Moderate to Severe Plaque Psoriasis: Pooled Results From Phase 2 and Phase 3 Randomized Clinical Trials. JAMA Dermatol. 2022 Jul 1;158(7):735-744. doi: 10.1001/jamadermatol.2022.1185. PMID 35544084

DOCUMENTS (1):
  • Informed Consent Form (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/58/NCT06338358/ICF_000.pdf